CLINICAL TRIAL: NCT02052986
Title: An Open-Label Study of Vascazen in Cardiac Rehab Patients With Deficient Blood Omega-3 Fatty Acid Levels
Acronym: CARE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: New York Hospital Queens (Other)
Collaborators: NYHQ Cardiac Health Center (Unknown); Pivotal Therapeutics (Unknown)
Responsible Party: Principal Investigator, Brian S. Marino, DO, Physician, New York Hospital Queens
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: VCT-01
Record Dates: First submitted 2013-12-16; First posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Dyslipidemia
Keywords: Fatty Acids, Omega-3; Omega-3 fatty acids; Docosahexaenoic acid (DHA); Eicosapentaenoic acid (EPA); Docosapentaenoic acid (DPA); Omega Index; Omega Score; Cardiac Rehab
MeSH Terms: conditions — Dyslipidemias | interventions — VASCAZEN

ARMS (1):
- Vascazen (Experimental): Enrolled patients will receive four capsules daily of VASCAZEN (a 3.0 gram daily dose of EPA+DHA) for a total of 12 weeks.
  Interventions: Other: VASCAZEN

INTERVENTIONS:
Other: VASCAZEN — All enrolled subjects will receive 4 capsules daily of VASCAZEN which delivers 3.0 grams of EPA and DHA

SUMMARY:
The investigators aim to test the hypothesis that dietary supplementation with VASCAZEN will correct omega-3 deficiency in cardiac rehab patients and improve biochemical risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (> or = 18 years of age)
* Enrolled in Cardiac Rehabilitation clinic with documented cardiovascular disease as assessed by the principle investigator
* Has had cardiovascular examination within the past 2 months

Exclusion Criteria:

* Subjects who refuse to provide written consent
* Subjects with medical conditions, as determined by the principal investigator, which prevented them from study participation
* Subjects with a known bleeding or clotting disorder
* Subjects with known allergies to fish
* Subjects with an implantable cardiac defibrillator
* Subjects with a heart transplant
* Female subjects who are currently taking hormone replacement therapy
* Subjects who are pregnant or planning on becoming pregnant
* Subjects currently taking Omega-3 fatty acid supplements (either under medical supervision or self-administered)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Change in sum of Omega-Score and Omega-Index | 12 weeks
  Change in the sum of the subject's blood Eicosapentaenoic acid (EPA) + Docosahexaenoic acid (DHA) + Docosapentaenoic acid (DPA) levels (Omega-Score) and the change in the sum of the subject's red blood cell (RBC) EPA + DHA levels (Omega-Index) over 12 weeks of study treatment with Vascazen

SECONDARY OUTCOMES:
Change in patient health questionnaire-9 (PHQ-9) depression scale | 12 weeks
  Change in patient health questionnaire-9 (PHQ-9) depression scale after 12 weeks of study treatment

OTHER OUTCOMES:
Change in Omega-3 Score and Omega-3 Index | Baseline, 6 weeks, 12 weeks
Change in high-sensitivity C-reactive protein (hsCRP) | Baseline, 6 weeks, 12 weeks
Change in blood levels of total cholesterol, low-density lipoprotein (LDL), high density lipoprotein (HDL), very-low density lipoprotein (VLDL) cholesterol and their subfractions (particle size) | Baseline, 6 weeks, 12 weeks
Change in blood level of Triglycerides | Baseline, 6 weeks, 12 weeks
Change in fasting plasma glucose | Baseline,12 weeks
Change in blood glucose and insulin measurements following administration of oral glucose tolerance test (OGTT) | Baseline, 12 weeks
Change in glycated hemoglobin (HbA1c) | Baseline,12 weeks
Change in Lipoprotein associated Phospholipase (Lp-PLA2) | Baseline, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian S Marino, DO, Principal Investigator — New York Hospital Queens
Locations (1):
- The NYHQ Cardiac Health Center, Fresh Meadows, New York, United States

REFERENCES:
- [Background] Albert CM, Campos H, Stampfer MJ, Ridker PM, Manson JE, Willett WC, Ma J. Blood levels of long-chain n-3 fatty acids and the risk of sudden death. N Engl J Med. 2002 Apr 11;346(15):1113-8. doi: 10.1056/NEJMoa012918. PMID 11948270
- [Background] Dietary supplementation with n-3 polyunsaturated fatty acids and vitamin E after myocardial infarction: results of the GISSI-Prevenzione trial. Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto miocardico. Lancet. 1999 Aug 7;354(9177):447-55. PMID 10465168
- [Background] Bays H. Clinical overview of Omacor: a concentrated formulation of omega-3 polyunsaturated fatty acids. Am J Cardiol. 2006 Aug 21;98(4A):71i-76i. doi: 10.1016/j.amjcard.2005.12.029. Epub 2006 May 30. PMID 16919519
- [Background] Mori TA, Burke V, Puddey IB, Watts GF, O'Neal DN, Best JD, Beilin LJ. Purified eicosapentaenoic and docosahexaenoic acids have differential effects on serum lipids and lipoproteins, LDL particle size, glucose, and insulin in mildly hyperlipidemic men. Am J Clin Nutr. 2000 May;71(5):1085-94. doi: 10.1093/ajcn/71.5.1085. PMID 10799369
- [Background] Grimsgaard S, Bonaa KH, Hansen JB, Nordoy A. Highly purified eicosapentaenoic acid and docosahexaenoic acid in humans have similar triacylglycerol-lowering effects but divergent effects on serum fatty acids. Am J Clin Nutr. 1997 Sep;66(3):649-59. doi: 10.1093/ajcn/66.3.649. PMID 9280188
- [Background] Geleijnse JM, Giltay EJ, Grobbee DE, Donders AR, Kok FJ. Blood pressure response to fish oil supplementation: metaregression analysis of randomized trials. J Hypertens. 2002 Aug;20(8):1493-9. doi: 10.1097/00004872-200208000-00010. PMID 12172309
- [Background] Thies F, Garry JM, Yaqoob P, Rerkasem K, Williams J, Shearman CP, Gallagher PJ, Calder PC, Grimble RF. Association of n-3 polyunsaturated fatty acids with stability of atherosclerotic plaques: a randomised controlled trial. Lancet. 2003 Feb 8;361(9356):477-85. doi: 10.1016/S0140-6736(03)12468-3. PMID 12583947
- [Background] Kris-Etherton PM, Harris WS, Appel LJ; American Heart Association. Nutrition Committee. Fish consumption, fish oil, omega-3 fatty acids, and cardiovascular disease. Circulation. 2002 Nov 19;106(21):2747-57. doi: 10.1161/01.cir.0000038493.65177.94. No abstract available. PMID 12438303
- [Background] Harris WS, Von Schacky C. The Omega-3 Index: a new risk factor for death from coronary heart disease? Prev Med. 2004 Jul;39(1):212-20. doi: 10.1016/j.ypmed.2004.02.030. PMID 15208005
- [Background] von Schacky C, Harris WS. Cardiovascular risk and the omega-3 index. J Cardiovasc Med (Hagerstown). 2007 Sep;8 Suppl 1:S46-9. doi: 10.2459/01.JCM.0000289273.87803.87. PMID 17876200
- [Background] Derosa G (2011) Effects of n-3 PUFA on Insulin Resistance After an Oral Fat Load. European Journal of Lipid Science. 113: (8) 950-960